CLINICAL TRIAL: NCT04356053
Title: Systematic Screening for Primary Immunodeficiencies in Patients Hospitalized for Severe Infections in Intensive Care : DIPREA
Brief Title: Systematic Screening for Primary Immunodeficiencies in Patients Hospitalized for Severe Infections in Intensive Care.
Acronym: DIPREA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0199
Record Dates: First submitted 2020-04-17; First posted 2020-04-22 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Primary Immunodeficiency
Keywords: severe infection; pediatric
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently about 90 cases of infection in children are reported every year in pediatric intensive care, a disease considered to be the main cause of hospitalization of children. 16% of invasive pneumococcal infections are linked to a genetic abnormality in immunity. Herpetic encephalitis has become a model of genetic infectious disease, with new mutations identified in the TLR3 pathway. Severe infections are no longer the result of chance and can be the way to reveal a primary immune deficiency. In this context, the investigators propose to evaluate the incidence of hereditary immune deficiency after a systematic immunological screening in children admitted for a severe infection in pediatric intensive care unit (ICU).

DETAILED DESCRIPTION:
Severe infection requiring admission in intensive care unit (ICU) are not so rare. A retrospective pilot study conducted at Montpellier University Hospital Center (UHC) between 2013 and 2015 showed that 19.7% of the pediatric ICU admissions were related to a severe infection. An isolated severe infectious episode could be related to a hereditary immune deficiency (HID), even though there are no history of recurrent clinical signs and biological stigmata. For example, Gaschignard and colleagues considered that 16% of the invasive pneumococcal infections are related to a genetic defect of immunity (doi: 10.1093/cid/ciu274). Growing evidence has shown that severe infectious diseases occurring in childhood are attributed to inborn errors of immunity (doi: 10.1073/pnas.1521651112). While the nosology of severe infections has strong links to inherited immune deficiency that are rare diseases affecting less than 1 birth / 5000, there are no prospective studies that assessed the incidence of primary immune deficiencies in children who presented a severe infection.

ELIGIBILITY:
Inclusion criteria:

* Subject aged 1 month to 16 years.
* Admission in pediatric ICU for more than 24h.
* Documented severe infection (bacterial, viral, fungal).
* Child benefiting from a social security scheme.
* Collection of parental consent / legal representatives.

Exclusion criteria:

* Prematurity (gestational age <37 weeks of gestation) up to 6 months of age.
* Undocumented severe infections.
* Children entered for isolated RSV bronchiolitis, with no other infectious related complications.
* Previous comorbidity explaining the infection and/or the stay in intensive care / continuous care: known primary or secondary immunodeficiency; burned; risk factors for status epilepticus (encephalopathy, known epilepsy, head trauma), pneumonia or asthma (swallowing disorders, tracheotomy, chronic pulmonary pathology, asthma), meningitis (cochlear implants, breccia, neuromeningeal material), deep infection (implanted material, recent surgery), cardiovascular decompensation.
* Any other chronic pathology favoring an infection
* Impossibility to obtain the consent of parents / legal representatives.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric population
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Immunological abnormalities | 1 day
  Immunological abnormalities : based on the screening test

SECONDARY OUTCOMES:
Diagnosis of primary immunodeficiency | 1 day
  Diagnosis of primary immunodeficiency

OTHER OUTCOMES:
duration of hospitalization | 1 day
  Compare the duration of hospitalization enter the group treated by alone antibiotic and the group treated by antibiotic and surgical drainage.

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle VIGUE, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC